CLINICAL TRIAL: NCT01223339
Title: A Phase 1, Randomized, Double Blind, Placebo-Controlled, Parallel Cohort, Single Dose Escalation And Multiple Dose Study In Japanese Healthy Subjects, And Open Label, Single Dose Escalation Study In Western Healthy Subjects To Investigate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of PF-04971729
Brief Title: Evaluation of Pharmacokinetics, Safety, And Tolerability Of Ertugliflozin (PF-04971729, MK-8835) In Japanese And Western Healthy Participants (MK-8835-041)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-041
Record Dates: First submitted 2010-10-13; First posted 2010-10-19 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Ertugliflozin; Japanese and Western population; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Dose Japanese Cohort (Experimental): This will be a single dose Cohort in which Japanese healthy participants will receive 3 ascending single doses (1 mg, 5 mg, and 25 mg) of ertugliflozin or placebo through 3 dosing periods. A minimum wash out period of 7-days will be set between each dose administration.
  Interventions: Drug: Ertugliflozin; Drug: Placebo
- Single dose Western cohort (Experimental): This will be a single dose Cohort in which Western healthy participants will receive 3 ascending single doses (1 mg, 5 mg, and 25 mg) of ertugliflozin through 3 dosing periods. A minimum wash out period of 7-days will be set between each dose administration.
  Interventions: Drug: Ertugliflozin
- Multiple Dose Japanese Cohort (Experimental): This will be a multiple dose Cohort in which Japanese healthy participants will receive once-daily 25 mg ertugliflozin or placebo for 7 days.
  Interventions: Drug: Ertugliflozin; Drug: Placebo

INTERVENTIONS:
Drug: Ertugliflozin — Dose escalation of 1, 5, and 25 mg Ertugliflozin administered in the fasted state
  Arms: Single Dose Japanese Cohort; Single dose Western cohort
Drug: Placebo — Placebo tablets to Ertugliflozin administered in the fasted state
  Arms: Single Dose Japanese Cohort
Drug: Ertugliflozin — Ertugliflozin 25 mg tablets administered once daily in the fed state for 7 days
  Arms: Multiple Dose Japanese Cohort
Drug: Placebo — Placebo tablets administered once daily in the fed state for 7 days
  Arms: Multiple Dose Japanese Cohort

SUMMARY:
This study is to characterize the pharmacokinetics, safety, tolerability, and pharmacodynamics of single and multiple oral doses (SD, MD) of ertugliflozin (PF-04971729, MK-8835) in Japanese healthy participants. The secondary objective is to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single doses of ertugliflozin in Western healthy participants as compared to Japanese healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential, between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Japanese subjects must have four Japanese grandparents who were born in Japan.
* Mean body weight and the body weight range of Western subjects are similar to those of Japanese subjects with a 10% plus and minus error.
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with scheduled visits, treatment plan,laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Asian or Polynesian subjects in Western subject groups.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males within 6 months of screening.
* History or evidence of habitual use of tobacco or nicotine containing products within 3 months of Screening, with the exception of light smoking (up to 5 cigarettes per day or the equivalent).
* Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 msec at screening.
* Subjects with ANY of the following abnormalities on safety laboratory tests):
* Evidence of glycosuria, as defined by a positive urine dipstick test;
* Fasting serum triglyceride >300 mg/dL;
* Fasting LDL-cholesterol > than or equal to 190 mg/dL.
* Fasting serum glucose >125 mg/dL.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of ertugliflozin for the Single Dose Cohort | Up to Day 4 of each treatment period
Time taken to reach the maximum observed plasma concentration (Tmax) of ertugliflozin for the Single Dose Cohort | Up to Day 4 of each treatment period
Area under the plasma concentration-time curve (AUC) from time 0 to time of the last quantifiable concentration (AUClast) for ertugliflozin for the Single Dose Cohort | Up to Day 4 of each treatment period
AUC from Hour 0 to infinity (AUCinf) for ertugliflozin for the Single Dose Cohort | Up to Day 4 of each treatment period
Ertugliflozin half life (t1/2) for the Single Dose Cohort | Up to Day 4 of each treatment period
Apparent clearance (CL/F) of ertugliflozin for the Single Dose Cohort | Up to Day 4 of each treatment period
Apparent volume of distribution (Vz/F) for the Single Dose Cohort | Up to Day 4 of each treatment period
Accumulation Ratio of Area Under the Curve for the dosing interval of ertugliflozin (Rac) for the Single Dose Cohort | Up to Day 4 of each treatment period
Number of participants who experienced an adverse event (AE) for the Single Dose Cohort | Up to 10 days after the final dose of study drug (Up to Day 11)
Number of participants who discontinued study drug due to an AE for the Single Dose Cohort | Up to Day 1 of each treatment period
Urinary Glucose Excretion over 24 hours for the Single Dose Cohort | Up to 24 hours postdose (Up to Day 2)
Cmax of ertugliflozin for the Multiple Dose Cohort | Up to Day 10
Tmax of ertugliflozin for the Multiple Dose Cohort | Up to Day 10
AUClast for ertugliflozin for the Multiple Dose Cohort | Up to Day 10
AUCinf for ertugliflozin for the Multiple Dose Cohort | Up to Day 10
t1/2 for the Multiple Dose Cohort | Up to Day 10
CL/F of ertugliflozin for the Multiple Dose Cohort | Up to Day 10
Vz/F for the Multiple Dose Cohort | Up to Day 10
Rac for the Single Dose Cohort | Up to Day 10
Number of participants who experienced an AE for the Multiple Dose Cohort | Up to 10 days after the final dose of study drug (Up to Day 17)
Number of participants who discontinued study drug due to an AE for the Multiple Dose Cohort | Up to Day 7
Urinary Glucose Excretion over 24 hours for the Multiple Dose Cohort | Up to 24 hours postdose (Up to Day 8)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819
- [Derived] Marshall JC, Liang Y, Sahasrabudhe V, Tensfeldt T, Fediuk DJ, Zhou S, Krishna R, Dawra VK, Wood LS, Sweeney K. Meta-Analysis of Noncompartmental Pharmacokinetic Parameters of Ertugliflozin to Evaluate Dose Proportionality and UGT1A9 Polymorphism Effect on Exposure. J Clin Pharmacol. 2021 Sep;61(9):1220-1231. doi: 10.1002/jcph.1866. Epub 2021 Jun 19. PMID 33813736
- [Derived] Li Y, Nucci G, Yamamoto Y, Fediuk DJ, Sahasrabudhe V. Pharmacokinetics and Pharmacodynamics of Ertugliflozin in Healthy Japanese and Western Subjects. Clin Pharmacol Drug Dev. 2021 Jul;10(7):765-776. doi: 10.1002/cpdd.908. Epub 2021 Jan 12. PMID 33434408